CLINICAL TRIAL: NCT07261293
Title: Effects of Blood Flow Restriction Aerobic Exercise on Systemic Inflammation, Hypoxia, Exercise Capacity, and Pulmonary Functions in Patients With Chronic Obstructive Pulmonary Disease: A Prospective Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction Aerobic Exercise on Inflammation, Hypoxia, Exercise Capacity, and Lung Function in COPD
Acronym: BFR-COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISTU-BFRAE-COPD25
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; BFR; Aerobic exercise; Exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Aerobic Exercise Group (Active Comparator): Participants in this group will perform low-intensity aerobic exercise on a cycle ergometer under blood flow restriction (BFR) as part of pulmonary rehabilitation. BFR pressure will be applied bilaterally to the proximal thighs using pneumatic cuffs at 40-50% of each participant's limb occlusion pressure. Sessions will include warm-up, 15 minutes of aerobic exercise, and cool-down, supervised by a physiotherapist. No aerobic exercise without BFR will be performed in this arm.
  Interventions: Behavioral: Blood Flow Restriction Aerobic Exercise Training
- Conventional Aerobic Exercise Group (Active Comparator): Participants in this arm will perform standard aerobic exercise on a cycle ergometer as part of conventional pulmonary rehabilitation without blood flow restriction. Exercise intensity will be prescribed at 60-80% of the target heart rate calculated using the Karvonen formula. Each session will include a 3-minute warm-up, 15 minutes of continuous aerobic exercise, and a 3-minute cool-down. Exercise intensity, frequency, and duration will be matched to the BFR aerobic exercise group. All sessions will be supervised by an experienced physiotherapist. No blood flow restriction will be applied in this arm.
  Interventions: Behavioral: Conventional Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Blood Flow Restriction Aerobic Exercise Training — Blood Flow Restriction Aerobic Exercise Training Participants will undergo aerobic exercise performed with blood flow restriction (BFR) applied to both thighs using pneumatic cuffs positioned at the proximal portion of the lower limbs. Cuff pressure will be individualized for each participant based on limb occlusion pressure (LOP), determined by Doppler assessment. During training, cuffs will be inflated to 40-50% of the participant's LOP and will remain inflated throughout the aerobic exercise phase. Sessions will include warm-up, continuous low-intensity cycling, and cool-down, supervised by a physiotherapist. The purpose of this intervention is to induce physiological adaptations associated with BFR, such as increased metabolic stress and muscular activation, while using low mechanical load.
  Arms: Blood Flow Restriction Aerobic Exercise Group
Behavioral: Conventional Aerobic Exercise Training — Participants in this group will perform aerobic exercise on a cycle ergometer without blood flow restriction (BFR) as part of standard pulmonary rehabilitation. The aerobic exercise protocol will be performed at 60-80% of the participant's target heart rate (THR), calculated using the Karvonen formula:
  THR = [(HRmax - HRrest) × % intensity] + HRrest.
  Training will be performed twice per week for a total of 8 weeks and will include 3 minutes of warm-up, 15 minutes of target-intensity aerobic cycling, and 3 minutes of cool-down (total duration: 21 minutes). Pedal resistance and cadence will be adjusted according to the Borg Rating of Perceived Exertion (RPE), with the target RPE maintained between 3 and 4. Exercise intensity (watt level) will be progressed weekly by approximately 5-10%, aligned with tolerance and RPE scores (Patterson et al., 2019). No BFR will be applied at any stage of the intervention.
  Arms: Conventional Aerobic Exercise Group

SUMMARY:
Purpose:

This study aims to compare the effects of the classical pulmonary rehabilitation (PR) program and blood flow restriction (BFR) applied during low-intensity aerobic exercise within PR on systemic inflammation, hypoxemia, exercise capacity, pulmonary function, respiratory muscle strength, and quality-of-life parameters in individuals with COPD.

Methods:

This randomized controlled study will include 34 individuals with COPD, allocated into a BFR aerobic group and a control group. Both groups will receive core PR components, including diaphragmatic breathing, pursed-lip breathing, respiratory muscle training, and peripheral muscle strengthening. The BFR group will perform low-intensity aerobic exercise with blood flow restriction, while the control group will perform moderate-intensity aerobic exercise without BFR in accordance with standard PR protocols. All sessions will be supervised by a physiotherapist, twice per week, for eight weeks. Systemic inflammation markers, arterial blood gases, pulmonary function, exercise capacity, quality of life, and symptom scores will be assessed before PR, after the 8th session, and at the end of the program. Data will be analyzed using SPSS 26.0.

Expected Contribution:

This study aims to provide evidence-based insights into the physiological and clinical effects of low-intensity BFR aerobic exercise within PR and to determine its potential advantages compared with classical PR. Additionally, it seeks to clarify whether low-intensity BFR aerobic exercise may serve as a better-tolerated alternative for COPD patients who experience exercise intolerance during moderate-intensity aerobic training.

DETAILED DESCRIPTION:
1. RATIONALE AND AIM OF THE STUDY

   Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory condition characterized by airflow limitation, systemic inflammation, impaired gas exchange, and significant skeletal muscle dysfunction. Individuals with COPD frequently experience reduced exercise capacity, peripheral muscle weakness, chronic hypoxemia, fatigue, sleep disturbances, and decreased quality of life. These systemic features contribute to increased symptom burden and diminished functional independence.

   Pulmonary rehabilitation (PR) is an established intervention that improves exercise tolerance, reduces dyspnea, and enhances quality of life. However, many patients are unable to sustain high-intensity exercise because of ventilatory limitations, early muscle fatigue, or oxygen desaturation. This creates a need for alternative exercise strategies that provide an adequate physiological stimulus while remaining tolerable for individuals with limited exercise reserve.

   Blood Flow Restriction (BFR) exercise is a low-intensity training method that induces localized hypoxic and metabolic stress, promoting physiological adaptations such as increased muscle activation and improved functional performance. Although early findings suggest potential benefits of BFR, its effects when integrated into a PR program-particularly on systemic inflammation, oxygenation, respiratory muscle function, and exercise capacity-have not been comprehensively investigated.

   This study aims to compare conventional PR with PR combined with low-intensity aerobic exercise performed under BFR in individuals with stable COPD. The study will evaluate systemic inflammatory markers, oxygenation and hypoxemia responses, exercise capacity, spirometric measurements, respiratory muscle strength, arterial blood gases, and patient-reported symptoms. By assessing physiological, functional, and subjective outcomes together, the study seeks to determine the potential added value of BFR-assisted aerobic training within pulmonary rehabilitation.

   The findings are expected to clarify whether BFR can enhance the effectiveness of PR, provide a more tolerable training option for individuals with limited exercise capacity, and support the development of individualized rehabilitation strategies for people with COPD.
2. DESIGN For this study, the sample will consist of patients aged 40-80 years with a diagnosis of COPD who are referred to the Pulmonary Rehabilitation Unit of the Department of Pulmonology at Sultan Abdülhamid Han Training and Research Hospital, University of Health Sciences, by a pulmonology specialist. Participants will be randomly assigned into two groups using a computerized randomization method: a routine pulmonary rehabilitation group (control group) and a group receiving blood flow restriction (BFR) during aerobic exercise, which is one of the parameters of pulmonary rehabilitation (intervention group). Pulmonary rehabilitation programs for both groups will be administered by an experienced physiotherapist under the supervision of a pulmonology specialist. Before initiating the rehabilitation program, the cardiovascular suitability of the patients for pulmonary rehabilitation will be determined by a cardiologist. The program will begin once medical approval indicating "suitable for pulmonary rehabilitation" has been obtained. The study has a multidisciplinary and multidimensional structure.

   Both groups will participate in a total of 16 pulmonary rehabilitation sessions conducted twice weekly for 8 weeks within the hospital. Each session will last 60 minutes.

   2.1. Intervention Group In the intervention group, the pulmonary rehabilitation program will include the active cycle of breathing techniques, diaphragmatic breathing, pursed-lip breathing, and respiratory muscle training. In addition, a bilateral resistance exercise program will be given to target the shoulder flexors, elbow flexors, and quadriceps muscle groups. Furthermore, aerobic exercise with blood flow restriction (BFR) will be performed on a cycle ergometer.

   Active Cycle of Breathing Techniques (ACBT) ACBT consists of a series of techniques applied to improve ventilation efficiency. These techniques strengthen respiratory muscles and enhance respiratory function. In this cycle, various breathing strategies are applied consecutively to increase ventilatory capacity. In COPD patients, these techniques help open the airways and optimize ventilation. Techniques include deep breathing, breath-holding, and controlled exhalation strategies.

   Diaphragmatic Breathing Diaphragmatic breathing is a method of inhalation performed using the diaphragm instead of the accessory muscles. This technique increases ventilation of the lower lungs, enhances oxygen uptake, and reduces respiratory muscle fatigue. In COPD patients, diaphragmatic breathing reduces the work of breathing and allows patients to breathe more efficiently.

   Pursed-Lip Breathing Pursed-lip breathing is a technique that helps keep the airways open during exhalation. The patient exhales slowly through lightly pursed lips during breathing. This technique facilitates overcoming airway resistance, regulates airflow in COPD patients, and enables more effective breathing. It also helps correct ventilation-perfusion imbalances and reduces dyspnea.

   Respiratory Muscle Training In this study, inspiratory muscle training will be performed using the Powerbreathe Medic Plus (gray) device twice a week for 8 weeks. The initial load will be set at 30% of the patient's measured maximal inspiratory pressure (MIP). Progression will be made according to the perceived difficulty level reported during exercise based on the Modified Borg Scale (0-10), keeping the perceived exertion (RPE) between 3-4 and increasing the load by 5-10% each week. The goal will be to reach 60% of the MIP. The training will follow a protocol of 5 breaths × 6 sets, with rest intervals adjusted based on patient tolerance.

   Peripheral Muscle Training Resistance training will be applied as 2 sets × 8 repetitions at an RPE of 3-4 on the Modified Borg Scale. Targeted muscle groups will include the quadriceps femoris, shoulder flexors, and elbow flexors.

   BFR + Aerobic Exercise Program BFR will be applied using a wireless AirBands cuff placed proximally on the thigh at the level of the femoral artery at 45% of the individual limb occlusion pressure (LOP). Aerobic exercise will be performed on a cycle ergometer at 40-60% of the target heart rate (low-moderate intensity). The target heart rate will be determined using the Karvonen formula [THR=HRmax-HRrest)×%intensite]+HRrest]. Each session will consist of 3 minutes of warm-up, 15 minutes of exercise, and 3 minutes of cool-down (21 minutes total). BFR will begin after warm-up and remain inflated throughout the exercise. At the end of the session, the cuff will be released, followed by a 5-minute reactive hyperemia period. Exercise progression will be individualized according to the MBS RPE scores recorded during each session; the target perceived effort will be kept between 2-3 (light-moderate), and workload (watts) will be increased by 5-10% weekly as tolerated.

   2.2. Control Group In the control group, the pulmonary rehabilitation program will include the active cycle of breathing techniques, diaphragmatic breathing, pursed-lip breathing, and respiratory muscle training. In addition, a bilateral resistance training program targeting the shoulder flexors, elbow flexors, and quadriceps muscle groups will be implemented. Aerobic exercise training will be performed on a cycle ergometer without the use of BFR.

   Active Cycle of Breathing Techniques (ACBT) ACBT consists of techniques applied to improve the efficiency of breathing. These techniques strengthen the respiratory muscles and enhance respiratory function. Various breathing strategies are applied consecutively to increase ventilatory capacity. In COPD patients, these strategies open the airways, optimize ventilation, and improve airflow. The cycle includes techniques such as deep breathing, breath-holding, and controlled exhalation.

   Diaphragmatic Breathing Diaphragmatic breathing is a method of breathing performed by effectively using the diaphragm rather than the abdominal or accessory muscles. This technique improves ventilation of the lower lungs, increases oxygen intake, and reduces respiratory muscle fatigue. In COPD patients, diaphragmatic breathing decreases the work of breathing and helps patients breathe more efficiently.

   Pursed-Lip Breathing Pursed-lip breathing is a technique that helps maintain airway patency during exhalation. The patient exhales slowly through lightly pursed lips. This technique facilitates overcoming airway resistance, regulates airflow in COPD patients, and makes breathing more efficient. It also corrects ventilation imbalances and reduces dyspnea.

   Respiratory Muscle Training Inspiratory muscle training will be performed using the Powerbreathe Medic Plus (gray) device, twice a week for 8 weeks. The initial training load will be set at 30% of the patient's measured maximal inspiratory pressure (MIP). Progression will be based on perceived exertion reported during exercise according to the Modified Borg Scale (0-10), maintaining an RPE of 3-4, with weekly increases of 5-10% in resistance. The goal is to reach 60% of the MIP. Training will follow the "5 breaths × 6 sets" format with individualized rest intervals according to patient tolerance.

   Peripheral Muscle Training Resistance training will be applied as 2 sets of 8 repetitions at an RPE of 3-4. Targeted muscle groups will include the quadriceps femoris, shoulder flexors, and elbow flexors.

   Aerobic Exercise Program The aerobic exercise protocol on the cycle ergometer will be performed at 60-80% of the target heart rate. The target heart rate will be calculated using the Karvonen formula, which incorporates the heart rate reserve (HRR):[THR=(HRmax-HRrest)×%intensite]+HRrest] This formula provides a more accurate estimation of the training heart rate, especially in clinical populations. Aerobic training will be performed twice weekly for 8 weeks, with each session consisting of 3 minutes of warm-up, 15 minutes of target aerobic exercise, and 3 minutes of cool-down (21 minutes total). Pedal resistance and pedaling speed will be adjusted according to the Borg RPE scores reported during the session. The target RPE during exercise will be kept at 3-4, with weekly increases of 5-10% in workload.
3. Sample Size Calculation

   The primary outcome of the study is the change in 6MWT distance. Based on previously reported clinically meaningful differences in 6MWT distance in individuals with COPD and assuming a medium effect size, a power analysis was performed using a significance level of 0.05 and a power of 80%. The calculation indicated that 17 participants per group (34 in total) would be sufficient to detect clinically relevant between-group differences in 6MWT distance.
4. Statistical Analysis

All data will be analyzed using a statistical software package. The normality of distribution for continuous variables will be assessed using appropriate tests. Parametric variables will be presented as mean ± standard deviation, and non-parametric variables as median with interquartile range.

Baseline differences between groups will be analyzed using independent samples t-tests or Mann-Whitney U tests, as appropriate. Categorical variables will be compared using the chi-square test.

Within-group changes from pre- to post-intervention will be evaluated using paired samples t-tests or Wilcoxon signed-rank tests, depending on data distribution. Group × time interactions will be examined using two-way repeated measures ANOVA or linear mixed models.

Correlations between changes in inflammatory markers and changes in 6MWT distance will be analyzed using appropriate correlation coefficients. A p-value of <0.05 will be considered statistically significant for all analyses, and effect sizes will be reported to aid interpretation of clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 40 and 80 years
* Clinically stable patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD) according to GOLD 2024 criteria with post-bronchodilator FEV₁/FVC < 0.70
* Stable clinical condition (no acute exacerbation within the past 4 weeks)
* Individuals clinically evaluated and approved as suitable for pulmonary rehabilitation (PR) participation by a cardiology specialist
* Functional capacity sufficient to participate in PR (e.g., 6-Minute Walk Test ≥150 m)
* No contraindications to blood flow restriction (BFR) training (e.g., no peripheral vascular disease, no active thrombosis)
* Ability to understand and follow instructions (adequate auditory and cognitive function)

Exclusion Criteria:

* Acute exacerbation of COPD, hospitalization, or systemic corticosteroid treatment within the past 4 weeks
* Severe cardiovascular disease (uncontrolled hypertension >180/110 mmHg, myocardial infarction within the past 6 months, unstable angina, congestive heart failure NYHA Class III-IV)
* Neurological or orthopedic conditions significantly limiting lower-extremity function (e.g., hemiplegia, amputation, severe osteoarthritis, knee prosthesis)
* Severe renal impairment (GFR <30 mL/min/1.73 m²) or severe hepatic failure
* History of lower-extremity surgery within the past 3 months
* Active malignancy or systemic infection
* Anemia or chronic inflammatory/autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease)
* History of venous thromboembolism
* Peripheral arterial disease
* Physician-diagnosed sarcopenia
* Psychiatric disorders (major depression, dementia, psychotic disorders) limiting adherence to the study protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Capacity | Baseline and 8 weeks after intervention
  Exercise capacity will be evaluated using the 6-Minute Walk Test (6MWT), conducted according to ATS guidelines in a 30-meter corridor. The total distance walked in 6 minutes (6MWD) will be recorded as the primary indicator of functional exercise capacity. The outcome measure will assess the change in 6MWT distance from baseline to 8 weeks following the intervention in COPD patients undergoing pulmonary rehabilitation with or without blood flow restriction (BFR). An increase in 6MWD reflects improvement in exercise capacity.

SECONDARY OUTCOMES:
Change in Systemic Inflammation (CRP Levels) | Baseline and 8 weeks after intervention
  Systemic inflammation will be assessed using serum C-reactive protein (CRP) levels. Blood samples will be collected at baseline and after the 8-week intervention. CRP concentration will be analyzed using standard laboratory biochemical methods. Changes in CRP levels will be used to evaluate the effect of the intervention on systemic inflammatory status.
Change in Systemic Inflammation (RDW Levels) | Baseline and 8 weeks after intervention
  Red cell distribution width (RDW), an inflammatory and hypoxia-related hematologic marker, will be measured using complete blood count analysis. RDW values obtained at baseline and after the 8-week intervention will be compared to evaluate changes in systemic inflammation.
Change in Arterial Oxygen Partial Pressure (PaO₂) | Baseline and 8 weeks after intervention
  Arterial oxygen partial pressure (PaO₂) will be measured using arterial blood gas analysis (ABG). Blood samples will be collected at baseline and after the 8-week intervention. PaO₂ values will be used to assess changes in arterial oxygenation and respiratory gas exchange following the intervention.
Change in Respiratory Function (FEV₁) | Baseline and 8 weeks after intervention
  Respiratory function will be assessed using forced expiratory volume in 1 second (FEV₁), measured via standardized spirometry following ATS/ERS guidelines. FEV₁ values will be recorded in liters and as a percentage of the predicted value. Measurements obtained at baseline and after the 8-week intervention will be compared to evaluate changes in pulmonary function.
Change in Respiratory Muscle Strength (MIP) | Baseline and 8 weeks after intervention
  Respiratory muscle strength will be assessed using maximal inspiratory pressure (MIP), measured with an electronic pressure manometer following ATS/ERS standards. MIP represents the maximum negative pressure generated during a forceful inspiratory effort against an occluded airway. Measurements obtained at baseline and after the 8-week intervention will be compared to evaluate changes in inspiratory muscle strength.

OTHER OUTCOMES:
Change in Peripheral Muscle Strength (Quadriceps Strength) | Baseline and 8 weeks after intervention
  Peripheral muscle strength will be assessed by measuring isometric quadriceps muscle force using a handheld digital dynamometer (Lafayette Manual Muscle Tester). Participants will perform maximal voluntary isometric contraction for 3-5 seconds in a standardized seated position. Three trials will be recorded with 30 seconds of rest between attempts, and the highest value (in Newtons) will be used for analysis. Measurements obtained at baseline and after the 8-week intervention will be compared to evaluate changes in quadriceps strength.
Change in Dyspnea (mMRC Score) | Baseline and 8 weeks after intervention
  Dyspnea severity will be assessed using the Modified Medical Research Council (mMRC) Dyspnea Scale, which rates perceived breathlessness from 0 (no dyspnea) to 4 (severe dyspnea during minimal activity). mMRC scores obtained at baseline and after the 8-week intervention will be compared to evaluate changes in dyspnea levels.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agustí, A., & Hogg, J. C. (2019). Update on the pathogenesis of chronic obstructive pulmonary disease. New England Journal of Medicine, 381(13), 1248-1256. Almeida, C. N. S., Fiel, J. A., Sarges, E. S. N. F., et al. (2020). Physiological response to the Glittre-ADL test in elderly COPD patients. Fisioterapia em Movimento, 33, e003322. Centner, C., et al. (2019). Low-load blood flow restriction training induces similar morphological and strength adaptations to high-load resistance training. Journal of Applied Physiology, 127(6), 1643-1655. Geddes, E. L., O'Brien, K., Reid, W. D., et al. (2008). Inspiratory muscle training in adults with chronic obstructive pulmonary disease: a systematic review. Respiratory Medicine, 102(12), 1715-1729. Global Initiative for Chronic Obstructive Lung Disease. (2024). Global strategy for the diagnosis, management, and prevention of COPD: 2024 Report. Gosselink, R., et al. (2011). Impact of inspiratory muscle training in patients with COPD: What is the evidence? European Respiratory Journal, 37(2), 416-425. Grønfeldt, B.M., Lindberg Nielsen, J., Mieritz, R.M., Lund, H. & Aagaard, P. (2020) Effect of blood-flow restricted vs heavy-load strength train ing on muscle strength: systematic review and meta-analysis. Scandinavian Journal of Medicine & Science in Sports, 30(5), 837-848. Guo, C. L., Sun, H. J., & Li, J. (2023). Neutrophil-to-lymphocyte ratio as a marker of COPD severity. Respiratory Medicine, 195, 106900. Hassan, A., & Jabbar, N. (2022). C-reactive protein as a predictor of severity in chronic obstructive pulmonary disease: An experience from a tertiary care hospital. Cureus, 14(8). Kohlbrenner, D., Kuhn, M., Manettas, A., Aregger, C., Peterer, M., Greco, N., ... & Clarenbach, C. (2024). Low-load blood flow restriction strength training in patients with COPD: a randomised single-blind pilot study. Thorax, 79(4), 340-348. Laghi, F., & Tobin, M. J. (2003). Disorders of the respiratory muscles. American Journal of Respirator